CLINICAL TRIAL: NCT01194037
Title: A Phase 1b/2a, Open-label,Randomized, Safety, Tolerability, Dose Finding, PK/PD, and Preliminary Efficacy Study of Subcutaneous Hanferon™ in Combination With Ribavirin in Treatment-naïve Subjects With Genotype 1 Hepatitis C
Brief Title: A Phase 1b/2a Study of SC Hanferon™ in Combination With Ribavirin in Treatment-naïve Subjects With Genotype 1 Hepatitis C
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: HanAll BioPharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HL-143IFN-SC-US-001
Record Dates: First submitted 2010-09-01; First posted 2010-09-02 (Estimated); Last update posted 2025-04-22 (Actual); Status verified 2014-02

CONDITIONS: Chronic Hepatitis C Infection; Genotype 1
Keywords: Hepatitis C; HCV; Interferon; Hanferon
MeSH Terms: conditions — Hepatitis C | interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Hanferon (low dose) sc weekly + ribavirin(RBV) oral daily (Experimental): Hanferon™ 30 μg SC weekly + ribavirin(RBV)1000 mg daily (body weight < 75kg) or ribavirin(RBV) 1200 mg daily (body weight ≥ 75 kg)
  Interventions: Drug: recombinant variant of interferon-alpha 2b; Drug: Ribavirin
- Hanferon (high dose) sc weekly + ribavirin(RBV) oral daily (Experimental): Hanferon™ 60 μg SC weekly + ribavirin(RBV) 1000 mg daily (body weight < 75kg) or ribavirin(RBV) 1200 mg daily (body weight ≥ 75 kg)
  Interventions: Drug: recombinant variant of interferon-alpha 2b; Drug: Ribavirin
- Pegasys 180 ug sc weekly + RBV oral daily (Active Comparator): Pegasys® 180 μg SC weekly + ribavirin(RBV) 1000 mg daily (body weight < 75kg) or ribavirin(RBV) 1200 mg daily (body weight ≥ 75 kg)
  Interventions: Drug: Peginterferon alfa-2a; Drug: Ribavirin

INTERVENTIONS:
Drug: recombinant variant of interferon-alpha 2b — SC, Weekly
  Other Names: Hanferon
  Arms: Hanferon (high dose) sc weekly + ribavirin(RBV) oral daily; Hanferon (low dose) sc weekly + ribavirin(RBV) oral daily
Drug: Peginterferon alfa-2a — SC Weekly
  Other Names: Pegasys
  Arms: Pegasys 180 ug sc weekly + RBV oral daily
Drug: Ribavirin — Oral administration (The daily dose of ribavirin(RBV) was 1000mg for subjects weighing < 75 kg or 1200 mg for subjects weighing ≥ 75 kg)

SUMMARY:
This is an open-label, randomized, safety, tolerability, dose-finding, PK/PD, and preliminary efficacy study of subcutaneous Hanferon™ in combination with ribavirin(RBV) in treatment-naïve subjects with genotype 1 hepatitis C.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the safety and tolerability of ascending doses of Hanferon™ in combination with ribavirin (RBV).

The secondary objective of this study is to define the PK and PD of ascending doses of Hanferon™ in combination with ribavirin(RBV). The exploratory objective of this study is to make a preliminary assessment of Hanferon™ efficacy in combination with ribavirin(RBV).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic hepatitis C genotype 1a or 1b
* Male or female aged 18 to 65 years, inclusive
* Compensated liver disease without evidence of cirrhosis
* No evidence of type 1 or 2 diabetes mellitus, lipodystrophy or polycystic ovary syndrome
* No history or presence of autoimmune or lymphoproliferative disease or hemoglobinopathies
* Stable medication doses for 1 month for the chronic disease if subjects have chronic diseases, including but not limited to hypertension and dyslipidemia

Exclusion Criteria:

* History of previous treatment of hepatitis C
* Currently use medication for psychiatric illness including depression, suicidal ideation, and psychosis
* History or presence of chronic liver disease
* History of drug or alcohol abuse within the past year
* Evidence of active illicit drug use
* Clinically significant abnormal electrocardiogram (ECG) or rhythm strip
* Female subject who has a positive urine pregnancy test or who is lactating

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-06-23 (Actual); Primary Completion 2011-11-28 (Actual); Study Completion 2011-11-28 (Actual)

PRIMARY OUTCOMES:
HCV RNA level | Week 4

SECONDARY OUTCOMES:
Proportion of patients who reach RVR | Week 4
PK & PD | Weeks 0 and 3

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Los Angeles, California
  - National City, California
  - Miami, Florida
  - Atlanta, Georgia
  - Lexington, Kentucky
  - New Orleans, Louisiana